CLINICAL TRIAL: NCT07001709
Title: The Effect of Abiraterone on the Metabolism of Oxycodone
Brief Title: Determining the Effect of Abiraterone on the Metabolism of Oxycodone in Men With Prostate Cancer (the ENABLE Study)
Acronym: ENABLE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Deventer Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ME23-42; 2023-505705-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-29; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Pain Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Cancer Pain | interventions — Oxycodone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Receive 15 mg oxycodone (direct release) without the use of abiraterone. The plasma concentration of oxycodone, noroxycodone, oxymorphone and noroxymorphone is measured. In addition, one blood sample is drawn for determine patient characteristics and genotyping of CYP3A4 and CYP2D6 is determined.
  Interventions: Drug: Oxycodone oral capsule 15 mg
- Abiraterone group (Other): Receive 15 mg oxycodone (direct release) and abiraterone. The plasma concentration of oxycodone, noroxycodone, oxymorphone and noroxymorphone is measured. In addition, one blood sample is drawn for determine patient characteristics, the serum through concentration of abiraterone and genotyping of CYP3A4 and CYP2D6 are determined.
  Interventions: Drug: Oxycodone oral capsule 15 mg; Drug: Abiraterone Acetate Tablets 500 mg

INTERVENTIONS:
Drug: Oxycodone oral capsule 15 mg — Single dose of 15 mg oxycodone direct release (both arm 1 and arm 2)
Drug: Abiraterone Acetate Tablets 500 mg — Abiraterone group: 1000 mg abiraterone acetate (at steady state)
  Arms: Abiraterone group

SUMMARY:
Prostate cancer often leads to bone metastases, which require adequate pain management with opioids such as oxycodone. This study investigates whether abiraterone - a drug used in the treatment of prostate cancer - affects the pharmacokinetics of oxycodone in order to improve pain management.

DETAILED DESCRIPTION:
Rationale: Oxycodone is an opioid receptor agonist metabolized primarily by CYP3A4, and to a lesser extent by CYP2D6. Abiraterone is an androgen biosynthesis inhibitor prescribed to men with castration resistant prostate cancer (CRPC). The ENABLE study is a follow-up to the ENZYME study in which it was described that enzalutamide increases oxycodone metabolism in patients with CRPC. It is expected that concomitant use of abiraterone has no clinically relevant effect on oxycodone's plasma concentration since it solely inhibits CYP2D6. Therefore, discontinuing abiraterone treatment is not expected to result in toxicity. This might positively affect pain management and pharmacovigilance in patients with CRPC.

Objective: To investigate the effect of abiraterone on the pharmacokinetics (PK) of oxycodone following a single dose of 15 mg normal-release oxycodone in men with prostate cancer.

Trial design: A prospective, open-label, two-arm parallel clinical study.

Subjects will visit the hospital once for approximately nine hours. After screening for hypercapnia, subjects will receive one oral dose of 15 mg (10 mg and 5 mg capsules) normal-release oxycodone. In total, nine blood samples will be collected during the day for the control group and ten blood samples for the abiraterone group. Seven blood samples will be collected at predetermined times (t= 0.5, 1, 1.5, 2, 3, 5, 8 hours) in order to analyze the metabolism of oxycodone. One blood sample will be collected to determine abiraterone serum trough concentrations (abiraterone arm). In addition, two blood samples will be collected for patient characteristics, including one sample for genotyping of CYP3A4 and CYP2D6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed prostate cancer;
* Males aged 18 years or older;
* Treated with abiraterone 1000 mg once daily for at least 10 days (abiraterone arm).
* Not treated with abiraterone 1000 mg once daily for at least 10 days (control arm).

Exclusion Criteria:

* Use of oxycodone short acting <48 hours, or long acting <96 hours prior to the study day;
* Use of other opioids in the 14 days prior to the study day (see also appendix A);
* Use of other medication that has pharmacokinetic or pharmacodynamics interactions with oxycodone (see also appendix A);
* Arm 1: dose reduction or successive days of treatment interruption within 10 days prior to the study day (arm 1);
* Arm 2: treatment with abiraterone within 10 days prior to the study day;
* A body mass index (BMI) outside the range of 18 - 30 kg/m2;
* If hypersensitive to oxycodone;
* patients suffering from diarrhea
* If any type of abnormality; active or symptomatic viral hepatitis or chronic liver disease (e.g. classification with Child-Pugh B, Child-Pugh C);
* Known metastases in the liver that would affect drug metabolism;
* Patients with a CYP3A4 or CYP2D6 polymorphism;
* Moderate-severe renal dysfunction (GFR <60 ml/min/1.73m2) that affects drug metabolism ;
* Subjects with significant respiratory depression resulting in the need of oxygen therapy or objective hypoventilation (respiratory rate <12/min);
* Hypercapnia (venous pCO2 outside the range of 5.5 - 6.7; pH outside the range 7.30 - 7.40);
* Subjects with, a history of bronchial asthma, chronic obstructive pulmonary disease or pulmonary heart disease;
* Subjects who started their first cycle of chemotherapy during the 2 weeks before the study day;
* Major surgery within 1 month prior to screening or planned surgery;
* A history of drug abuse
* Patients receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine) and/or suffering from opioid withdrawal
* Patients with evidence of clinically significant gastrointestinal disease;
* Patients who are contraindicated for blood sampling;
* Unable to swallow solid, oral dosage forms whole with water;
* Participation in a clinical trial study at the time of enrolment or within 30 days or 5 half-lives of enrolment, whichever is longer;
* Previous gastric bypass or gastric band surgery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with prostate cancer
Enrollment: 29 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cmax Oxycodone | Measured at one of the time points (t= 0.5, 1, 1.5, 2, 3, 5, 8 hours)
  Maximum measured concentration of oxycodone
T1/2 oxycodone | t= 0.5, 1, 1.5, 2, 3, 5, 8 hours
  Measured half-life of oxycodone
AUC0-8h oxycodone | From 0 to 8 hours after ingestion of oxycodone
  Area under the curve of oxycodone from 0 to 8 hours after ingestion of oxycodone.

SECONDARY OUTCOMES:
Cmax noroxycodone | Measured at one of the time points (t= 0.5, 1, 1.5, 2, 3, 5, 8 hours)
  Maximum measured concentration of noroxycodone
AUC0-8h noroxycodone | From 0 to 8 hours after ingestion of oxycodone
  Area under the curve of noroxycodone from 0 to 8 hours after ingestion of oxycodone.
Cmax oxymorphone | Measured at one of the time points (t= 0.5, 1, 1.5, 2, 3, 5, 8 hours)
  Maximum measured concentration of oxymorphone
AUC0-8h oxymorphone | From 0 to 8 hours after ingestion of oxycodone
  Area under the curve of oxymorphone from 0 to 8 hours after ingestion of oxycodone.
Cmax noroxymorphone | Measured at one of the time points (t= 0.5, 1, 1.5, 2, 3, 5, 8 hours)
  Maximum measured concentration of noroxymorphone
AUC0-8h noroxymorphone | From 0 to 8 hours after ingestion of oxycodone
  Area under the curve of noroxycodone from 0 to 8 hours after ingestion of oxycodone.

CONTACTS AND LOCATIONS:
Locations (1):
- Deventer Ziekenhuis, Deventer, Overijssel, Netherlands